CLINICAL TRIAL: NCT00995267
Title: The Influence of the Family as Agents of Change on Eating Habits and Obesity in First and Second Grade School Children in Israel.
Brief Title: Eating Habits and Obesity in First and Second Grade School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LBoo1-HMO-CTIL
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2009-10

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; nutrition; exercise; Alfred Adler; schoolchildren; intervention study; community-based trial; parent-child interaction; nutritional behaviors
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- behavioral intervention (Experimental): Behavioral intervention arm comprises 5 joint parent-child school-based nutritional activities in which nutritional information was combined with Adler's behavioral concepts. and a 5-session parental workshop.
  Interventions: Behavioral: parent-child interaction/activities based on Adler's methods
- control arm (No Intervention)

INTERVENTIONS:
Behavioral: parent-child interaction/activities based on Adler's methods — Description of the Intervention:
  5 joint classroom activities (parents and children together, involving children in food choices/food preparation-sense of belonging/decision making): 1. Healthy breakfasts and 10 o'clock snacks 2. Fats and oils in the diet, cooking methods, setting limits to oily food intake. 3. Fruit and vegetables in the daily diet, adults as role models. 4. Learning about food categories & pyramid, healthy eating and growth. 5. Limiting consumption of sweets and snacks.
  Workshop for Parents: Explaining nutritional needs of children; how to encourage good eating habits, how to deal with children's manipulations, providing tools to elicit change; use of food to attract parental attention; practical tools to deal with their children's eating habits/obesity/refusal to eat/chronic health problems/failure to grow; ways to prevent use of food as an answer to childhood frustrations.
  Arms: behavioral intervention

SUMMARY:
Purpose: In the framework of a randomized concurrent controlled trial, to assess the effectiveness of a feasible educational mechanism based on the principles of Alfred Adler, that focuses on the family, to improve the dietary habits of schoolchildren, to induce them to increase their physical activity, and to prevent obesity and diseases related to obesity. Primary Objectives for Children: 1.To increase intake of fruits and vegetables, to reduce intake of sweets and unhealthy snacks at home and in school, to increase exercise and to reduce sedentary activities. Primary Objective for the Parents: Increase the involvement of parents in the education of their children regarding nutrition.

Description: Study population: Approximately 600 students and 600 parents from 24 first grade classes in 4 schools. Schools are randomized into intervention and control groups. The intervention comprises a 5-session parental workshop and 5 joint parent-child school-based activities. The control group will be offered the intervention after conclusion of the trial.

Participants are recruited in first grade, anthropometrics are measured, and pupils and parents are interviewed on eating habits and exercise. Snacks are observed. The intervention takes place in the second grade, and outcome assessment is done at the end of the 2nd grade and beginning of the 3rd grade. In-depth interviews will be conducted with parents of obese children.

Significance: Most interventions geared to prevention of childhood obesity have failed dismally. A new approach that focuses on the parent-child interaction may be contributory.

DETAILED DESCRIPTION:
Of the 743 children in 23 2nd grade classes in 4 schools, parents provided informed consent for 508 (68%), and again for 432 (58%) at the 3rd grade follow-up.

First stage of Recruiting 2007-2008: 3 first grade in each of 4 schools participating in the study. Total 12 classes. After the recruitment, initial data collection was conducted.

2008-2009: Allocation of students in 2nd grade from cycle 1 to intervention and control groups. Intervention in the experimental group. Data collection at the beginning and end of second grade. Recruiting new first grade classes (cycle 2), Primary data collection was conducted.

2009-2010: Completion of the follow-up cycle I. Last data collection at the beginning of the third grade. Allocation students 2nd grade from cycle 2 for intervention or control groups. Intervention in the experimental group of cycle 2. Data collection at the beginning and end of the second grade.

2010-2011: End of follow-up cycle 2. Collect data at the beginning of the third grade.

Description of the Intervention:

1. 5 joint parent-child classroom activities on the subject of nutrition, undertaken separately in the 12 intervention classes of the 4 clusters (ie. 60 sessions).
2. 5 workshops based on the approach of Adler that were restricted to parents, undertaken separately in the evenings for the 12 intervention classes (ie 60 sessions).

The control group (11 classes) had no intervention, but was identically monitored from first through third grade.

ELIGIBILITY:
Inclusion Criteria:

* All children in regular first grade classes in 4 schools whose parents provided informed consent

Exclusion Criteria:

* Schools with separate classes for boys and girls, and schools/classes for children with special needs

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 508 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome: change in intake of fruits, vegetables, sweets and unhealthy snacks at home, and exercise (questionnaire-based); and observed intake in school snacks | first grade to third grade

SECONDARY OUTCOMES:
change in BMI and waist circumference | first grade to third grade

CONTACTS AND LOCATIONS:
Overall Officials: Tori Goldstein, MSC, Principal Investigator — Hebew University Faculty of Medicine; Jeremy D Kark, MD PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel